CLINICAL TRIAL: NCT05745857
Title: A Phase 2 Intervention Study: Detection of Early Esophageal Neoplastic Lesions by Quantified Fluorescence Molecular Endoscopy Using Oral and Topical Administration of Bevacizumab-800CW and Cetuximab-800CW
Brief Title: Oral Bevacizumab-800CW and Cetuximab-800CW Administration to Detect Early Esophageal Adenocarcinomas
Acronym: SLURP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, dr. W.B. Nagengast, MD, Prof. Dr., University Medical Center Groningen
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 16054
Record Dates: First submitted 2023-02-02; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Barrett's Esophagus Without Dysplasia; Barrett Oesophagitis With Dysplasia; Esophageal Adenocarcinoma
Keywords: Fluorescence molecular endoscopy; Spectroscopy; Barrett's esophagus; Esophageal adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Barrett Esophagus | interventions — Bevacizumab; Cetuximab; Spectrum Analysis

STUDY DESIGN:
Intervention Model Description: Arm 1: Oral bevacizumab-800CW If oral administration is feasible the investigators will move on to arm 2, if it does not seem feasible the investigators will move on to arm 3.
  Arm 2: Oral cetuximab-800CW The investigators will move on to combined oral bevacizumab-800CW/cetuximab-800CW if oral cetuximab-800CW seems feasible. If it does not seem feasible, they will administer oral bevacizumab-800CW to a control group of non-dysplastic Barrett's esophagus patients.
  Arm 3 (only performed if oral administration does not work) Topical administration of bevacizumab-800CW compared to combined topical administration of bevacizumab-800CW/cetuximab-800CW. This group will be expanded if combined administration increases lesion detection. If this is not the case, the investigators will include a control group of non-dysplastic patients with Barrett's esophagus as a control group who will receive topical bevacizumab-800CW.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral bevacizumab-800CW (Experimental): Dose finding of oral bevacizumab-800CW and extend optimal dose group (n = 5 - 10)
  Interventions: Drug: Avastin; Device: Fluorescence endoscopy and multi-diameter single fiber reflectance/single fiber fluorescence (MDSFR/SFF) spectroscopy
- Oral cetuximab-800CW and combined oral cetuximab-800CW and bevacizumab-800CW (Experimental): Dose finding of oral cetuximab-800CW in first five patients and combined oral bevacizumab-800CW and cetuximab-800CW if the investigators see good results with cetuximab-800CW. If not, they will add a control group of non-dysplastic BE patients and administer oral bevacizumab-800CW.
  (n = 15)
  Interventions: Drug: Avastin; Drug: Erbitux; Device: Fluorescence endoscopy and multi-diameter single fiber reflectance/single fiber fluorescence (MDSFR/SFF) spectroscopy
- Combined topical tracer administration bevacizumab-800CW and cetuximab-800CW (Experimental): This arm will only be part of the study when oral administration is not feasible or safe.
  Compare single topical tracer administration of bevacizumab-800CW with combined topical tracer administration of bevacizumab-800CW and cetuximab-800CW. Extend combined group when lesion detection is increased or add control group with non-dysplastic BE patients if not.
  (n = 20)
  Interventions: Drug: Avastin; Drug: Erbitux; Device: Fluorescence endoscopy and multi-diameter single fiber reflectance/single fiber fluorescence (MDSFR/SFF) spectroscopy

INTERVENTIONS:
Drug: Avastin — Orally administered
  Other Names: Bevacizumab
Drug: Erbitux — Orally administered
  Other Names: Cetuximab
  Arms: Combined topical tracer administration bevacizumab-800CW and cetuximab-800CW; Oral cetuximab-800CW and combined oral cetuximab-800CW and bevacizumab-800CW
Device: Fluorescence endoscopy and multi-diameter single fiber reflectance/single fiber fluorescence (MDSFR/SFF) spectroscopy — Fluorescent endoscope fiber and spectroscopy probe will be inserted through the working channel of the normal clinical therapeutic endoscope

SUMMARY:
Previous studies have confirmed the great potential of quantitative fluorescence molecular endoscopy (qFME) when looking at additional lesion detection initially missed by high-definition white light endoscopy (HD-WLE) for surveillance of Barrett's esophagus.

DETAILED DESCRIPTION:
However, the investigators hypothesized, that additional lesions can potentially be identified by simultaneous use of two targeted tracers because of variable expression of vascular endothelial growth factor A (VEGFA) and epidermal growth factor receptor (EGFR )within oesophageal adenocarcinoma (EAC). Until now, solely intravenous and topical administration of the tracers has been investigated. However, optimization of tracer administration and shortened incubation is necessary for clinical translation and implementation of this new technique from Barrett's esophagus (BE) expert centers to regional non-expert centers. BE surveillance procedures normally takes up to 15 minutes at regional hospitals, of which most of the procedural time is needed to take biopsies according to the Seattle protocol. Introducing qFME into these hospitals would elongate the procedure time with at least 10 - 15 minutes. This would increase healthcare costs and put increased pressure on BE healthcare. Ideally, the gastroenterologist can immediately start with the qFME procedure without any incubation time while maintaining the best target-to-background ratios (TBR) possible. Oral administration by drinking the tracer prior to the procedure would eliminate incubation time and its consequences. Quantified qFME with oral tracer administration and targeted biopsies could potentially replace the time-consuming, high miss rate Seattle protocol, improve lesion detection and decrease global healthcare costs associated with BE.

ELIGIBILITY:
Inclusion Criteria:

* BE patients without dysplasia and with suspected/diagnosed low-grade dysplasia (LGD), high-grade dysplasia (HGD) or superficial EAC and planned diagnostic and/or therapeutic endoscopy
* Written informed consent is obtained

Exclusion Criteria:

* Patients under the age of eighteen.
* Submucosal and invasive EAC, also defined as EAC with tumor, node and metastasis (TNM)-classification other than T1.
* Previous radiation therapy for esophageal cancer
* Known immunoglobulin allergy
* Previous chemotherapy, immunotherapy or related surgery
* Prior bevacizumab or cetuximab treatment
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of shortening qFME procedural time by oral administration of bevacizumab-800CW and cetuximab-800CW for the detection of BE neoplasia. | 12 months
  Evaluating the performance of qFME with oral administration of bevacizumab-800CW and cetuximab-800CW for detection of neoplasia in BE patients compared to HD-WLE. This comparison will be based on target-to-background rations calculated from the in vivo fluorescence images and quantified by MDSFR/SFF spectroscopy measurements
Evaluate if the combination of tracers improves lesion detection by the number of invisible lesions detected | 12 months
  Increased lesion detection in % compared to previously gathered amount of invisible lesions with topical tracer administration

SECONDARY OUTCOMES:
Collect safety data on oral administration of (combined) bevacizumab-800CW and cetuximab-800CW. | Five minutes before and ten minutes after tracer administration
  Blood pressure in millimeters of mercury (mmHg)
Heart rate | Five minutes before and ten minutes after tracer administration
  Beats per minute
Temperature | Five minutes before and ten minutes after tracer administration
  Degrees Celsius
To (semi)quantify and evaluate the in vivo fluorescent signal of bevacizumab-800CW and cetuximab-800CW | 12 months
  Correlate and validate fluorescence signals detected in vivo with ex vivo histopathology grade of dysplasia and VEGFA and EGFR expression
Eventually further specify and objectify the improvement of qFME by standardisation | 12 months
  Determining optimal pre-set features for gain and exposure times for our fluorescence camera system

CONTACTS AND LOCATIONS:
Overall Officials: Wouter B. Nagengast, Prof. dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No